CLINICAL TRIAL: NCT00777595
Title: A Randomized, Double Blind, Single Dose, Positive and Placebo Controlled, Crossover Study of the Effects of Inhaled Carmoterol, at the Proposed Therapeutic and Supratherapeutic Doses, on the QTc Intervals in Healthy Subjects
Brief Title: Evaluation of Possible Effects on the QTc Interval of CHF 4226 pMDI in Healthy Volunteers
Acronym: CT14
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Steven E. Linberg, Ph.D., Chiesi Pharmaceuticals Inc.
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCD-0808-PR-0036
Record Dates: First submitted 2008-10-20; First posted 2008-10-22 (Estimated); Last update posted 2009-03-27 (Estimated); Status verified 2009-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: QTc; CHF 4226 HFA; pMDI; Carmoterol
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment A (Experimental): Single therapeutic dose of CHF 4226 pMDI
  Interventions: Drug: CHF 4226 pMDI
- Treatment B (Experimental): Single supratherapeutic dose of CHF 4226 pMDI
  Interventions: Drug: CHF 4226 pMDI
- Treatment C (Placebo Comparator): Single dose of placebo
  Interventions: Drug: Placebo
- Treatment D (Active Comparator): Single dose of moxifloxacin
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: CHF 4226 pMDI — Inhaled solution, single therapeutic dose
  Other Names: Carmoterol HFA
  Arms: Treatment A
Drug: CHF 4226 pMDI — Inhaled solution, single supratherapeutic dose
  Other Names: Carmoterol HFA
  Arms: Treatment B
Drug: Placebo — Inhaled solution, single dose of placebo
  Arms: Treatment C
Drug: Moxifloxacin — Tablet, oral, 400mg, single dose
  Other Names: Avelox
  Arms: Treatment D

SUMMARY:
The purpose of this study is to evaluate the effect of single doses of therapeutic and supratherapeutic doses of inhaled CHF 4226 pMDI on ventricular repolarization in healthy subjects compared with placebo.

DETAILED DESCRIPTION:
The secondary purposes of this study are to 1) determine if there is a relationship between the duration of the QTc intervals and the plasma concentrations of carmoterol; 2) expand the available information on plasma pharmacokinetics and urine excretion for inhaled carmoterol at the proposed therapeutic and supra-therapeutic doses; and 3) generate additional safety information.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male or female subjects, 18-55 years of age who provided written informed consent.
* A body mass index (BMI) between 18 - 30, inclusive.
* A normal blood pressure (< 140mmHg systolic and < 90mmHg diastolic)
* A normal 12-lead ECG (QTcF interval < 450msec for males and < 470msec for females).
* A serum potassium </= 4.0mEq/L.
* A calculated creatinine clearance > 80mL/min.
* Male subjects must agree to use a medically acceptable contraceptive (abstain from sexual intercourse, or use a condom with spermicide), have had a vasectomy at least 6 months prior to study participation or have a partner who is not of childbearing potential.

Exclusion Criteria:

* A history or presence of significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease.
* A history of sensitivity or allergy to the quinolone class of antibiotics and/or a beta 2 adrenergic receptor agonist.
* Clinically significant screening results (laboratory profiles, medical histories, ECGs, physical exam).
* Hemoglobin below the normal reference range for the testing laboratory.
* Abuse of alcohol or other substances.
* Current use of tobacco products.
* Subjects with a positive laboratory test result for hepatitis B, hepatitis C, HIV, controlled substances, cotinine or alcohol.
* Any prescription medication taken within 14 days (or 5 elimination half-lives, whichever is longer) of Study Day -2, or have taken any over-the-counter medications, including topical medications, vitamins, herbal or dietary supplements/remedies (e.g., Saint John's Wort or Milk Thistle), within 14 days of Study Day -2, or planned concomitant medication while in the study (except for acetaminophen up to 2g/day), with the exception of hormonal birth control medications or hormone replacement therapy for females.
* A history of additional risk factors for Torsade de Pointes (e.g., hypokalemia, history of drowning survival, family history of Long QT Syndrome, family history of Short QT Syndrome, or family history of unexplainable early sudden death).
* Subject is pregnant or lactating female, or female at risk of pregnancy (i.e., not using an adequate contraceptive method: surgical sterilization [e.g., bilateral tubal ligation], hormonal contraception [implantable, patch, oral], IUD, and double-barrier methods [any double combination of: male or female condom with spermicidal gel, diaphragm, sponge, cervical dap]_.
* Participation in a study of an investigational drug within 30 days prior to the baseline ECG.
* Any condition that, in the judgment of the Investigator, would place a subject at undue risk, or potentially compromise the results or interpretation of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2008-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
QTci | ECGs taken every treatment period on day -1 and day +1 at -1, -0.5, -0.25, 0.08, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hrs

SECONDARY OUTCOMES:
QTcX interval (subject-specific correction of QTcF, QTcB and QTcH) | ECGs taken every treatment period on day -1 and day +1 at -1, -0.5, -0.25, 0.08, 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hrs
Plasma concentration (AUC, Cmax, Tmax) | Each treatment period on dosing day at -0.75, 0.08, 0.25, 0.5, 1, 2, 4, 6, 8 and 12 hrs
Urinary excretion (Ae) | Each treatment period on day of dosing at -0.75, 0.58 and 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Robert I. Cooper, MD, Principal Investigator — PRACS Institute, Ltd.; Steven E. Linberg, PhD, Study Director — Chiesi Farmaceutici S.p.A.
Locations (1):
- PRACS Institute, Ltd., Fargo, North Dakota, United States

REFERENCES:
- [Background] Russell T, Riley SP, Cook JA, Lalonde RL. A perspective on the use of concentration-QT modeling in drug development. J Clin Pharmacol. 2008 Jan;48(1):9-12. doi: 10.1177/0091270007311115. No abstract available. PMID 18094215
- [Background] Garnett CE, Beasley N, Bhattaram VA, Jadhav PR, Madabushi R, Stockbridge N, Tornoe CW, Wang Y, Zhu H, Gobburu JV. Concentration-QT relationships play a key role in the evaluation of proarrhythmic risk during regulatory review. J Clin Pharmacol. 2008 Jan;48(1):13-8. doi: 10.1177/0091270007307881. PMID 18094216
- [Background] Bloomfield D, Krishna R. Commentary on the clinical relevance of concentration/QTc relationships for new drug candidates. J Clin Pharmacol. 2008 Jan;48(1):6-8. doi: 10.1177/0091270007312257. No abstract available. PMID 18094214